CLINICAL TRIAL: NCT03816020
Title: NAD-PARK: A Double-blinded Randomized Pilot Trial of NAD-supplementation in Drug naïve Parkinson's Disease
Brief Title: NAD-supplementation in Drug naïve Parkinson's Disease
Acronym: NAD-PARK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2018/597
Record Dates: First submitted 2018-12-07; First posted 2019-01-25 (Actual); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Parkinson Disease; Neurodegenerative Diseases
Keywords: clinical pilot, Nicotamide Riboside, Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases | interventions — nicotinamide-beta-riboside

STUDY DESIGN:
Intervention Model Description: After initial assessment at baseline, the participants will be randomly assigned (1:1) to one of two study groups (n = 15 per group): NR 500 mg x 2/day, or placebo. Participants and investigators will be masked to treatment group.
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants and investigators will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NR Group (Active Comparator): Participants receiving Nicotinamide Riboside capsules, 500mg BI'D for 30 days
  Interventions: Dietary Supplement: Nicotinamide Riboside
- Placebo Group (Placebo Comparator): Participant receiving Placebo BIDfor 30 days
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Nicotinamide Riboside — Nicotinamide Riboside capsules 250mg x 2 BID
  Arms: NR Group
Other: Placebo — Placebo capsules BID
  Arms: Placebo Group

SUMMARY:
1. Primary objective: Determine if NR has an impact on the neurometabolic profile of patients with PD as measured by [18F]Fluorodeoxyglucose (FDG)-positron emission tomography (FDG-PET).
2. Secondary objective: Determine whether high dose oral NR improves motor symptoms associated with PD.
3. Tertiary objectives: determine whether high dose oral NR rectifies NAD metabolism and increases NAD levels in body fluids and muscle tissue.

DETAILED DESCRIPTION:
Individuals with PD (n=30) will be recruited starting 14/02/2019 from the department of Neurology, Haukeland University Hospital. Only newly diagnosed and drug naïve PD patients are eligible for inclusion. After initial assessment at baseline, the participants will be randomly assigned (1:1) to one of two study groups (n = 15 per group): Nicotamide Riboside (NR) 500 mg x 2/day, or placebo. Participants and investigators will be masked to treatment group. Participants and investigators will be blinded (double blinded). The study will have a 4 week exposure period, during which patients will self-administer NR 500 mg x 2/day, or placebo per os. Patients will not be using any dopaminergic treatment during the study period. During baseline and 4 week follow-up, MDS-UPDRS will be performed as clinical measure. We will also collect blood, cerebral spinal fluid and muscle biopsy from all subjects at baseline and 4 week follow-up. Imaging will be performed using MRI, DAT Scan and FDG-PET at baseline and 4 week follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed with PD
2. Drug naïve with respect to dopaminergic treatment
3. Have a clinical diagnosis of idiopathic PD according to the MDS clinical diagnostic criteria for PD

Exclusion Criteria:

1. [¹²³I]FP-CIT single photon emission CT (DaTscan) does not show nigrostriatal degeneration.
2. Magnetic resonance imaging (MRI) suggestive of atypical parkinsonsism.
3. Dementia or other neurological disorder at baseline visit
4. Metabolic, neoplastic, or other physically or mentally debilitating disorder at baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-03-09 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
PDRP changes from NR use | 4 weeks
  The primary outcome will be the between-group difference in Parkinson's disease related pattern (PDRP) measured by FDG-PET comparing baseline and 3-4 week follow-up measurement.

SECONDARY OUTCOMES:
Motoric change of symptoms from NR use | 4 weeks
  Clinical changes measured by MDS-UPDRS from using NR

OTHER OUTCOMES:
Determine whether high dose oral NR rectifies NAD metabolism in body fluids and muscle tissue. | 4 weeks
  To measure NAD a liquid chromatography/tandem mass spectrometry will be use (abrv platform for method is LC-MS/MS.) We are interested in change of value of NAD. There is to our knowledge no measured NAD levels of PD patients. See PMID: 29184669 for the same method that we will use.

CONTACTS AND LOCATIONS:
Overall Officials: Charalampos Tzoulis, PhD, Principal Investigator — Nevro-Sysmed
Locations (1):
- Haukeland University Hospital, Bergen, Hordaland, Norway

IPD SHARING:
Plan to Share IPD: No
Data will only be shared if there is scientific collaboration. Will not be publicaly shared.

REFERENCES:
- [Derived] Brakedal B, Dolle C, Riemer F, Ma Y, Nido GS, Skeie GO, Craven AR, Schwarzlmuller T, Brekke N, Diab J, Sverkeli L, Skjeie V, Varhaug K, Tysnes OB, Peng S, Haugarvoll K, Ziegler M, Gruner R, Eidelberg D, Tzoulis C. The NADPARK study: A randomized phase I trial of nicotinamide riboside supplementation in Parkinson's disease. Cell Metab. 2022 Mar 1;34(3):396-407.e6. doi: 10.1016/j.cmet.2022.02.001. PMID 35235774